CLINICAL TRIAL: NCT05409391
Title: Study to Assess the Efficacy and Safety of Insulin Titration System Based on Deep Learning on Glucose Control in Type 2 Diabetes Mellitus Patients
Brief Title: Insulin Titration System Based on Deep Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoying Li, Professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSE-202205
Record Dates: First submitted 2022-06-01; First posted 2022-06-08 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus Type 2 - Insulin-Treated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI (Experimental): Insulin Titration System Based on Deep Learning
  Interventions: Device: Insulin Titration System

INTERVENTIONS:
Device: Insulin Titration System — A noval insulin titration system, which is based on deep learning

SUMMARY:
This is an open-labeled, one-arm intervention trial to access the effect and safety of the Insulin Titration System Based on Deep Learning in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The study enrolls 13 patients with Type 2 Diabetes in Zhongshan Hospital who are on treatment with insulin. After screening for the inclusion and exclusion criteria, eligible patients will receive insulin dosage titration set by the Insulin Titration System Based on Deep Learning in the intervention trial. The goal of insulin therapy was to achieve preprandial capillary blood glucose between 5.6-7.8 mmol/L and postprandial capillary glucose less than 10.0mmol/L. All patients are studied for 5 consecutive days or untill hospital discharge. For each patient, capillary glucose concentration was measured at 7 time points of fasting, after breakfast, before and after lunch, before and after dinner, and before bedtime a day using Glucometer (Glupad, Sinomedisite, China). Capillary glucose measurements were performed by the nurse staff according to standard procedures with a point-of-care testing device, which is integrated into the HIS system. And continuous glucose monitoring (CGM) was performed using flash glucose monitoring (Abbott Freestyle Libre, USA) placed on the upper left arm. This study will be conducted in the Department of Endocrinology, Zhongshan Hospital,Fudan University.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* age of 18-75 years
* HbA1c between 7.0% and 11.0%.

Exclusion Criteria:

* subjects with acute complications of diabetes, such as ketoacidosis or hyperglycemic hyperosmolar state;
* BMI ≥ 45kg/m2;
* women who are pregnant or breast-feeding;
* subjects with severe cardiac, hepatic, renal diseases; subjects with any psychiatric or psychological diseases;
* subjects with severe edema, infections or peripheral circulation disorders, receiving surgery during hospitalization;
* subjects who could not comply with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
mean daily blood glucose concentration | 5 days
  For each patient, capillary glucose concentration was measured at 7 time points of fasting, after breakfast, before and after lunch, before and after dinner, and before bedtime a day using Glucometer (Glupad, Sinomedisite, China). Capillary glucose measurements were performed by the nurse staff according to standard procedures with a point-of-care testing device, which is integrated into the HIS system. The primary outcome is the difference in glycemia control as measured by mean daily blood glucose concentration during the intervention period.

SECONDARY OUTCOMES:
glucose concentration in target range (TIR) of 3.9-10.0 mmol/L | 5 days
  TIR measured by CGM and Capillary glucose measurements, respectively
glucose concentration above range (10.1-13.9 mmol/L or >13.9 mmol/L) | 5 days
  TAR measured by CGM and Capillary glucose measurements, respectively
glucose concentration below range (3.0-3.8 mmol/L or <3.0 mmol/L) | 5 days
  TBR measured by CGM and Capillary glucose measurements, respectively
glycemic variability | 5 days
  glycemic variability measured by CGM and Capillary glucose measurements, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Department of Endocrinology, Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang G, Liu X, Ying Z, Yang G, Chen Z, Liu Z, Zhang M, Yan H, Lu Y, Gao Y, Xue K, Li X, Chen Y. Optimized glycemic control of type 2 diabetes with reinforcement learning: a proof-of-concept trial. Nat Med. 2023 Oct;29(10):2633-2642. doi: 10.1038/s41591-023-02552-9. Epub 2023 Sep 14. PMID 37710000